CLINICAL TRIAL: NCT06766019
Title: Adebrelimab Combined With Irinotecan Liposomal (II), Oxaliplatin, and 5-FU/LV Conversion Therapy for Locally Advanced Pancreatic Cancer: a Prospective, Single-arm, Exploratory Clinical Study
Brief Title: Adebrelimab Combined With Irinotecan Liposomal (II), Oxaliplatin, and 5-FU/LV Conversion Therapy for Locally Advanced Pancreatic Cancer
Status: Active, not recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: PC-IIT-003
Record Dates: First submitted 2025-01-05; First posted 2025-01-09 (Actual); Last update posted 2025-01-09 (Actual); Status verified 2025-01

CONDITIONS: Pancreatic Cancer
Keywords: Locally advanced pancreatic cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — irinotecan sucrosofate; Oxaliplatin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Adebrelimab combined with irinotecan liposomal (II), oxaliplatin, and 5-FU/LV (Experimental): Adebrelimab combined with irinotecan liposomal (II), oxaliplatin, and 5-FU/LV
  Interventions: Drug: Adebrelimab combined with irinotecan liposomal (II), oxaliplatin, and 5-FU/LV

INTERVENTIONS:
Drug: Adebrelimab combined with irinotecan liposomal (II), oxaliplatin, and 5-FU/LV — 1. adebrelimab 1200mg, i.v. D1, q28d
  2. irinotecan liposomal (II) 60mg/m^2, i.v. D1, Q2W
  3. oxaliplatin 85mg/m^2, i.v. D1, Q2W
  4. 5-FU/LV 2400mg/400mg/m^2, i.v. D1, Q2W 4-week cycles, 6 cycles

SUMMARY:
This trial is a prospective, single-arm, single-center, phase II clinical study, mainly targeting subjects with locally advanced pancreatic cancer, to explore the efficacy and safety of adebrelimab combined with irinotecan liposome (II), oxaliplatin, and 5-FU/LV conversion in the treatment of locally advanced pancreatic cancer.

DETAILED DESCRIPTION:
Subjects enter the screening period after being fully informed and signing an informed consent form. The screening period for the study is 28 days.

After completing the screening inspection and evaluation, patients will receive adebrelimab once and irinotecan liposomal (II), oxaliplatin, 5-FU/LV twice per cycle (4 weeks), and imaging of tumor lesions will be performed every 2 cycles (8 weeks ± 7 days) to evaluate whether patients can undergo surgery until surgical resection, disease progression, or intolerable toxicity, start of new anticancer drug therapy, withdrawal from the study, death, or loss to follow-up.

After 6 cycles of treatment, patients who are assessed to have no progression but are still unable to undergo radical surgical resection will receive maintenance treatment regimen (using capecitabine or teggio plus adebrelimab), and imaging efficacy will be evaluated every 12 weeks (± 7 days) during maintenance treatment. Surgical resectability will still be evaluated during maintenance treatment until disease progression or intolerable toxicity, start of new anticancer drug treatment, withdrawal from the study, death, or loss to follow-up.

ELIGIBILITY:
Inclusion Criteria:

-

Patients must meet all of the following inclusion criteria to be enrolled in this trial:

1. Sign written informed consent before implementing any trial-related procedures;
2. Age ≥ 18 years old and ≤ 70 years old, regardless of gender;
3. Locally advanced pancreatic cancer confirmed by histopathological/cytopathological examination;
4. Patients with locally advanced stage and no previous anti-tumor treatment (radiotherapy, chemotherapy, targeted or immunotherapy, etc.);

   Definition of locally advanced pancreatic cancer:
   1. The tumor has no distant metastasis;
   2. Pancreatic head/uncinate process: the tumor contacts the superior mesenteric artery > 180 ˚;
   3. Body and tail of pancreas: the tumor contacts the superior mesenteric artery or trunk celiac artery > 180 ˚; The tumor contacted the celiac trunk artery and infiltrated the abdominal aorta;
   4. The tumor invaded the jejunal branch of the superior mesenteric artery. The portal vein-superior mesenteric vein cannot be safely reconstructed due to tumor invasion, venous occlusion or involvement of a large area of the jejunal branch of the superior mesenteric vein;
5. According to the efficacy evaluation criteria of solid tumors (RECIST version 1.1) with at least one radiographically measurable lesion;
6. ECOG score 0-1;
7. If the biliary obstruction needs to be lifted, the expected survival time is > 3 months;
8. Sufficient organ function, subjects must meet the following laboratory indicators:

   1. Absolute neutrophil value (ANC) ≥ 1.5 × 109/L in the absence of granulocyte colony-stimulating factor in the past 14 days;
   2. platelets ≥ 100 × 109/L in the absence of blood transfusion in the past 14 days;
   3. hemoglobin > 9 g/dL in the absence of blood transfusion or use of erythropoietin in the past 14 days;
   4. total bilirubin ≤ 1.5 × upper limit of normal (ULN);
   5. aspartate aminotransferase (AST) and alanine aminotransferase (ALT) are ≤ 2.5 × ULN;
   6. blood creatinine ≤ 1.5 × ULN and creatinine clearance (calculated using the Cockcroft-Gault formula) ≥ 60 mL/min;
   7. Good coagulation function, defined as International Normalized Ratio (INR) or Prothrombin Time (PT) ≤ 1.5 times the ULN;
   8. euthyroidism, defined as thyroid stimulating hormone (TSH) within the normal range. If the baseline TSH is outside the normal range, subjects with total T3 (or FT3) and FT4 within the normal range can also be enrolled;
9. For female subjects of childbearing age, a negative urine or serum pregnancy test should be performed within 3 days prior to the first dose of study drug (Cycle 1, Day 1). If the urine pregnancy test result cannot be confirmed as negative, a blood pregnancy test is ordered. Women of non-childbearing age are defined as at least 1 year after menopause, or have undergone surgical sterilization or hysterectomy;
10. If there is a risk of conception, all subjects (whether male or female) are required to use contraception with an annual failure rate of less than 1% throughout the entire treatment period until 120 days after the last dose of study drug (or 180 days after the last dose of chemotherapy drug).

Exclusion Criteria:

-

Subjects who meet any of the following criteria will not be allowed to enter the study:

1. Patients with portal hypertension or cavernous degeneration of portal vein; Patients with gastrointestinal bleeding caused by tumors that have involved the gastrointestinal tract; Patients with tumor involvement of digestive tract causing intra-abdominal fistula or abscess; The tumor surrounds the celiac trunk or superior mesenteric artery (SMA) and causes significant involvement of the vascular wall (worm-like changes); Presence of distant metastatic lesions;
2. There is a third space effusion that cannot be controlled by drainage or other methods (such as medium-massive pleural effusion, medium-massive pericardial effusion, ascites); A small amount of pleural effusion or ascites that has no clinical symptoms and does not require clinical intervention should be strictly controlled before enrollment;
3. Those with poor compliance and inability to cooperate and describe treatment responses;
4. Other malignant diseases other than pancreatic cancer diagnosed within 5 years before the first dose (excluding radical basal cell carcinoma of the skin, squamous cell carcinoma of the skin, and/or radical resection of carcinoma in situ);
5. Currently participating in interventional clinical study treatment, or received other study drugs or treatment with study devices within 4 weeks prior to the first dose;
6. Have previously received the following therapies: anti-PD-1, anti-PD-L1, or anti-PD-L2 drugs or drugs directed at another stimulation or synergistic inhibition of T cell receptors (e.g., CTLA-4, OX-40, CD137);
7. Have received systemic systemic treatment with ready-for-use traditional Chinese medicine or immunomodulatory drugs with anti-tumor indications (including thymosin, interferon, interleukin, except for local use to control ascites) within 2 weeks before the first dose;
8. Active autoimmune disease requiring systemic therapy (e.g., use of disease-modifying drugs, glucocorticoids, or immunosuppressants) within 2 years prior to the first dose. Replacement therapy (e.g. thyroxine, insulin, or physiological glucocorticoids for adrenal or pituitary insufficiency, etc.) is not considered systemic therapy;
9. Were receiving systemic glucocorticoid therapy (excluding nasal spray, inhalation, or other routes of topical glucocorticoids) or any other form of immunosuppressive therapy within 7 days prior to the first dose of the study; Note: Physiological doses of glucocorticoids (≤ 10 mg/d of prednisone or equivalent) are allowed;
10. Known allogeneic organ transplantation (except corneal transplantation) or allogeneic hematopoietic stem cell transplantation;
11. Those who are known to be allergic to the active ingredients or excipients of the study drug adebelimab, leucovorin, 5-fluorouracil, irinotecan and oxaliplatin;
12. have not sufficiently recovered from any intervention-induced toxicities and/or complications prior to initiation of treatment (toxicities that have not been resolved by prior antineoplastic therapy, defined as not resolved to the level specified in the National Cancer Institute Common Terminology Criteria for Adverse Events ((NCI CTCAE v5.0) Grade 0 or 1, or inclusion/exclusion criteria, Except for hair loss/pigmentation. For subjects with irreversible toxicity that is not expected to worsen after study drug administration (e.g. hearing loss), enrollment will be determined at the discretion of the investigator);
13. People who are addicted to bad drugs such as drug abuse, long-term alcoholics, and people with infectious diseases such as AIDS (i.e. HIV 1/2 antibody positive);
14. Uncontrolled active hepatitis B (defined as HBsAg positive and detected HBV-DNA copy number greater than the upper limit of normal value in the laboratory of the study center);

Note: Subjects with hepatitis B who meet the following criteria can also be enrolled:

1. HBV viral load < 1000 copies/mL (200 IU/mL) prior to the first dose, subjects should receive anti-HBV therapy to avoid viral reactivation throughout the study drug treatment period;
2. For subjects with anti-HBc (+), HBsAg (-), anti-HBs (-), and HBV viral load (-), prophylactic anti-HBV therapy is not required, but close monitoring for viral reactivation is required; (15) Active HCV-infected subjects (HCV antibody positive and HCV-RNA levels above the lower detection limit); (16) Live vaccination within 30 days prior to the first dose (Cycle 1, Day 1); Note: Injectable inactivated viral vaccine against seasonal influenza is allowed up to 30 days prior to the first dose; However, it is not allowed to receive live attenuated influenza vaccine administered intranasally.

(17) pregnant or breastfeeding women; (18) Presence of any serious or uncontrollable systemic disease, such as:

1. The resting electrocardiogram has major abnormalities in rhythm, conduction or morphology with severe symptoms that are difficult to control, such as complete left bundle branch block, heart block above degree II, ventricular arrhythmia or atrial fibrillation;
2. Unstable angina pectoris, congestive heart failure, and chronic heart failure with New York Heart Association (NYHA) grade ≥ 2;
3. Any arterial thrombosis, embolism or ischemia, such as myocardial infarction, unstable angina pectoris, cerebrovascular accident or transient ischemic attack, has occurred within 6 months before enrollment for treatment;
4. Unsatisfactory blood pressure control (systolic blood pressure > 140 mmHg, diastolic blood pressure > 90 mmHg);
5. History of non-infectious pneumonia requiring glucocorticoid therapy within 1 year prior to the first dose, or current clinically active interstitial lung disease;
6. active pulmonary tuberculosis;
7. the presence of an active or uncontrolled infection requiring systemic treatment;
8. Clinically active diverticulitis, abdominal abscess, and gastrointestinal obstruction;
9. liver diseases such as cirrhosis, decompensated liver disease, acute or chronic active hepatitis;
10. Urine routine suggests urine protein ≥ + +, and 24-hour urine protein quantification > 1.0 g is confirmed;
11. Those who have mental disorders and are unable to cooperate with treatment;

(19) Medical history or disease evidence that may interfere with the results of the trial, prevent the subject from participating in the whole study, abnormal treatment or laboratory test values, or other situations that the investigator believes are not suitable for enrollment. The investigator believes that there are other potential risks that the investigator is not suitable for participating in this study.

Ages: 18 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 47 (Estimated)
Dates: Start 2024-10-16 (Actual); Primary Completion 2027-09-30 (Estimated); Study Completion 2027-09-30 (Estimated)

PRIMARY OUTCOMES:
Surgical conversion rate | Up to 6 months
  Refers to the proportion of subjects with successful conversion to all subjects receiving conversion therapy. Achievement of R0/R1 resection after conversion therapy was defined as successful conversion.

SECONDARY OUTCOMES:
Overall Survival (OS) | 5 years
  Time from start of patient treatment to death from any cause
1-year OS rate | 1 year
  Proportion of subjects who have survived 1 year from the date of first treatment after enrollment to all treated subjects
Objective response rate (ORR) | Up to 3 years
  Proportion of subjects including complete response (CR) or partial response (PR)
Event-free survival (EFS) | Up to 3 years
  The EFS endpoint is a composite time-to-event endpoint, and the "treatment failure" event is defined as the earliest occurrence of the following events: a. Failure to achieve local disease-free status after completion of conversion therapy and/or surgery (i.e., failed resection or disease progression resulting in inoperability); b. Local or distant recurrence; c. Death;
Disease Control Rate (DCR) | Up to 3 years
  Proportion of subjects whose best response observed throughout the study was CR, PR, or stable disease (SD)
Duration of response (DoR) | Up to 3 years
  From the first tumor response (CR or PR) to disease progression (PD) or death (whichever occurs earlier)
Time to disease progression (TTP) | Up to 3 years
  The time from the date of enrollment to the first observation of PD

OTHER OUTCOMES:
Treatment-related adverse events | Up to 3 years
  Observe all patients for any adverse events during the clinical study, including abnormalities in clinical symptoms and vital signs, abnormalities in laboratory tests, record their clinical manifestation characteristics, severity, time of occurrence, duration, treatment methods and prognosis, and determine their correlation with the investigational drug.
CA19-9 Response Rate | Up to 3 years
  Tumor marker response rates were assessed by changes in CA19-9 serum concentrations. Tumor marker response was defined as at least one concentration reduction of at least 50% from baseline occurring during the course of treatment. Only subjects with baseline values greater than the upper detection limit will be included in the evaluation of tumor marker response.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital with Nanjing Medical University, Nanjing, Jiangsu, China

IPD SHARING:
Plan to Share IPD: No